CLINICAL TRIAL: NCT02713529
Title: A Phase1b/2 Study Assessing Safety and Anti-tumor Activity of AMG 820 in Combination With Pembrolizumab in Select Advanced Solid Tumors
Brief Title: Safety and Efficacy Study of AMG 820 and Pembrolizumab Combination in Select Advanced Solid Tumor Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AmMax Bio, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150195; MASTERKEY (Other: Amgen); 2016-001080-36 (EudraCT Number); KEYNOTE-347 (Other: Merck)
Record Dates: First submitted 2016-03-03; First posted 2016-03-18 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Colorectal Cancer; Non-Small Cell Lung Cancer
Keywords: Solid Tumor; Pancreatic Cancer; Colorectal Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG820 and pembrolizumab (Experimental): Treatment with AMG820 and pembrolizumab
  Interventions: Biological: AMG820 and pembrolizumab

INTERVENTIONS:
Biological: AMG820 and pembrolizumab — Treatment with AMG820 and pembrolizumab

SUMMARY:
A multi-center Phase 1b/2 study testing the combination of AMG 820 and pembrolizumab in subjects with select advanced solid tumors.

DETAILED DESCRIPTION:
Phase 1b is AMG 820 dose determining and aimed at assessing the safety and tolerability of the selected starting dose of AMG 820 in combination with pembrolizumab. Phase 2 of the study will further evaluate safety and tolerability and additionally test whether AMG 820 can enhance the anti-tumor activity observed historically with pembrolizumab alone and/or overcome lack of response to pembrolizumab monotherapy in subjects with select solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, advanced colorectal, pancreatic or non-small cell lung cancer that is refractory to standard treatment, or the subjects have been intolerant to or refuse standard treatment.
* Measurable disease per RECIST 1.1 guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Adequate hematologic, renal, and hepatic function determined by laboratory blood and urine tests.
* Availability of recent tumor tissue within 3 months prior to enrollment, when feasible.

Exclusion Criteria:

* Has known active central nervous system metastases and/or carcinomatous meningitis.
* History of other malignancy with the past 2 years with some exceptions
* Evidence of active non-infectious pneumonitis/interstitial lung disease
* Evidence of other active autoimmune disease that has required prolonged systemic treatment in past 2 years.
* Evidence of clinically significant immunosuppression such as organ or stem cell transplantation, any severe congenital or acquired cellular and/or humoral immune deficiency, concurrent opportunistic infection.
* Receiving systemic immunostimulatory agents within 6 weeks or 5 half-lives, whichever is shorter, prior to first dose of study treatment (except ant PD-1/PD-L1 treatment if recruited into Group 4a or 4b).
* Evidence of active infection within 2 weeks prior to first dose of study treatment.
* Prior chemotherapy, radiotherapy, biological cancer therapy or major surgery within 28 days prior to enrollment
* Currently participating or has participated in a study (treatment period only) of an investigational agent or used an investigational device within 28 days of enrollment
* Received live vaccine within 28 days prior to enrollment
* Adverse event due to cancer therapy administered more than 28 days prior to enrollment that has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better.
* Positive for human immunodeficiency virus (HIV), Hepatitis B or C
* Women planning to become pregnant or who are lactating/breastfeeding while on study through 4 months after receiving the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (7):
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Australia (2):
  - Research Site, Camperdown, New South Wales
  - Research Site, Parkville, Victoria
- Research Site, Wilrijk, Belgium
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Research Site, Heidelberg, Germany
- Research Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Razak AR, Cleary JM, Moreno V, Boyer M, Calvo Aller E, Edenfield W, Tie J, Harvey RD, Rutten A, Shah MA, Olszanski AJ, Jager D, Lakhani N, Ryan DP, Rasmussen E, Juan G, Wong H, Soman N, Smit MD, Nagorsen D, Papadopoulos KP. Safety and efficacy of AMG 820, an anti-colony-stimulating factor 1 receptor antibody, in combination with pembrolizumab in adults with advanced solid tumors. J Immunother Cancer. 2020 Oct;8(2):e001006. doi: 10.1136/jitc-2020-001006. PMID 33046621
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 15 centers in Australia, Canada, United States of America, and Europe.
Pre-assignment Details: Part 1 was a phase Ib safety study comprised of two cohorts. Part 2 was a phase 2 safety and efficacy study comprised of 5 groups.
Groups:
- Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg: Part 1 Cohort 2 includes participants with advanced solid tumors who were treated with 1100 mg AMG 820 plus 200 mg pembrolizumab (Pem) every three weeks (Q3W) to determine safety. Participants could be treated up to 24 months if treatment was tolerable and clinical benefit was observed.
- Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg: Part 1 Cohort 1 includes participants with advanced solid tumors who were treated with 1400 mg AMG 820 plus 200 mg pembrolizumab (Pem) every three weeks (Q3W) to determine safety. Participants could be treated up to 24 months if treatment was tolerable and clinical benefit was observed.
  If >= 3 participants had dose limiting toxicities (DLTs), a second cohort was created with a lower AMG 820 dose + Pem 200 mg.
- Part 2, Group 1: CRC MMR-proficient: Group 1 is comprised of participants with colorectal cancer (CRC) who are proficient in mismatch repair genes (MMR).
  AMG 820 was administered at the recommended dose of 1100 mg intravenously in combination with pembrolizumab 200 mg every 3 weeks (± 3 days). Each group in Part 2 was evaluated separately using a Simon 2-stage design. Treatment continued until confirmed disease progression per modified irRECIST, or intolerance of study treatment, or clinically significant deterioration of health status requiring discontinuation, whichever occurred first, or the subject withdrew consent.
- Part 2, Group 2: Pancreatic Cancer: Group 2 is comprised of participants with advanced pancreatic cancer who are naïve to anti programmed-death 1 (PD-1), anti PD-ligand 1 (PD-L1), colony stimulating factor 1 (CSF-1) and colony stimulating factor 1 receptor (CSF-1R) therapies.
  AMG 820 was administered at the recommended dose of 1100 mg intravenously in combination with pembrolizumab 200 mg every 3 weeks (± 3 days). Each group in Part 2 was evaluated separately using a Simon 2-stage design. Treatment continued until confirmed disease progression per modified irRECIST, or intolerance of study treatment, or clinically significant deterioration of health status requiring discontinuation, whichever occurred first, or the subject withdrew consent.
- Part 2, Group 3: NSCLC PD-L1 Low, Naïve: Group 3 is comprised of participants with non-small cell lung cancer (NSCLC) who have low (< 50%) tumor PD-L1- expression and are naïve to anti-PD-1/PD-L1/CSF-1/CSF-1R agents.
  AMG 820 was administered at the recommended dose of 1100 mg intravenously in combination with pembrolizumab 200 mg every 3 weeks (± 3 days). Each group in Part 2 was evaluated separately using a Simon 2-stage design. Treatment continued until confirmed disease progression per modified irRECIST, or intolerance of study treatment, or clinically significant deterioration of health status requiring discontinuation, whichever occurred first, or the subject withdrew consent.
- Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low: Group 4a is comprised of participants who did not respond to or who relapsed during monotherapy with anti-PD-1/PD-L1 agents and are anti-CSF-1/CSF-1R naïve. These participants have low PD-L1 tumor expression (<50%).
  AMG 820 was administered at the recommended dose of 1100 mg intravenously in combination with pembrolizumab 200 mg every 3 weeks (± 3 days). Each group in Part 2 was evaluated separately using a Simon 2-stage design. Treatment continued until confirmed disease progression per modified irRECIST, or intolerance of study treatment, or clinically significant deterioration of health status requiring discontinuation, whichever occurred first, or the subject withdrew consent.
- Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High: Group 4b is comprised of participants who did not respond to or who relapsed during monotherapy with anti-PD-1/PD-L1 agents and are anti-CSF-1/CSF-1R naïve. These participants have high PD-L1 tumor expression (>=50%).
  AMG 820 was administered at the recommended dose of 1100 mg intravenously in combination with pembrolizumab 200 mg every 3 weeks (± 3 days). Each group in Part 2 was evaluated separately using a Simon 2-stage design. Treatment continued until confirmed disease progression per modified irRECIST, or intolerance of study treatment, or clinically significant deterioration of health status requiring discontinuation, whichever occurred first, or the subject withdrew consent.
Period: Overall Study
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Started | 8 | 7 | 42 | 31 | 4 | 19 | 6
Completed | 1 | 3 | 11 | 2 | 1 | 5 | 2
Not Completed | 7 | 4 | 31 | 29 | 3 | 14 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 3 | 26 | 27 | 3 | 13 | 3

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High | Total
Number analyzed (Participants) | 8 | 7 | 42 | 31 | 4 | 19 | 6 | 117
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 2 | 6 | 24 | 18 | 3 | 7 | 4 | 64
  65-74 years | 6 | 1 | 15 | 10 | 1 | 6 | 2 | 41
  75-84 years | 0 | 0 | 3 | 3 | 0 | 5 | 0 | 11
  >=85 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 16 | 14 | 1 | 1 | 3 | 43
  Male | 3 | 4 | 26 | 17 | 3 | 18 | 3 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 8 | 6 | 36 | 29 | 4 | 19 | 6 | 108
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4
  White | 8 | 5 | 39 | 26 | 4 | 17 | 5 | 104
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0 | 6 | 4 | 19 | 7 | 1 | 4 | 2 | 43
    Grade 1 | 2 | 3 | 23 | 24 | 3 | 15 | 4 | 74
    Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Number of Prior Line of Therapy [Count of Participants; unit: Participants]
  0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 9
  2 | 1 | 1 | 9 | 13 | 1 | 7 | 3 | 35
  3 | 4 | 3 | 11 | 8 | 0 | 7 | 3 | 36
  4 | 1 | 1 | 10 | 5 | 0 | 1 | 0 | 18
  5 | 2 | 2 | 10 | 2 | 0 | 3 | 0 | 19
  >5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease Stage at Screening [Count of Participants; unit: Participants] — There are five stages of cancer: stage 0 (or, carcinoma in situ), stage I, stage II, stage III, and stage IV. Lower stages indicate that the disease is more localized, or contained, whereas higher stages refer to cancers that have spread into other areas of the body.
  Participants
    Stage I | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Stage II | 1 | 0 | 3 | 3 | 1 | 1 | 0 | 9
    Stage III | 0 | 0 | 4 | 2 | 0 | 2 | 1 | 9
    Stage IV | 6 | 6 | 35 | 26 | 3 | 16 | 5 | 97

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicities (DLT)
Description: DLTs were evaluated by the Dose Level Review Team (DLRT). A DLT was defined as any grade >=3 adverse event occurring during a DLT time window (21 day period from the initial administration of AMG 820 and pembrolizumab in combination), and if judged by the investigator to be related to the administration of AMG 820 and/or pembrolizumab.
Time Frame: The DLT evaluation period was Day 1 to Day 21
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 8 | 7 | 41 | 31 | 4 | 19 | 6
Participants
  Participants with treatment emergent DLTs | 0 | 1 | 3 | 2 | 0 | 1 | 0
  DLT: Autoimmune pancreatitis | 0 | 1 | 0 | 0 | 0 | 0 | 0
  DLT: Autoimmune hepatitis | 0 | 1 | 0 | 0 | 0 | 0 | 0
  DLT: Cholecystitis | 0 | 1 | 0 | 0 | 0 | 0 | 0
  DLT: Electrolyte imbalance | 0 | 1 | 0 | 0 | 0 | 0 | 0
  DLT: Fatigue | 0 | 0 | 1 | 0 | 0 | 0 | 0
  DLT: Aspartate aminotransferase increased | 0 | 0 | 1 | 1 | 0 | 0 | 0
  DLT: Lipase increased | 0 | 0 | 0 | 0 | 0 | 1 | 0
  DLT: Epilepsy | 0 | 0 | 0 | 1 | 0 | 0 | 0
  DLT: Rash generalised | 0 | 0 | 1 | 0 | 0 | 0 | 0
  DLT: Rash maculo-papular | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Participants With Treatment -Emergent Adverse Events (TEAEs)
Description: TEAEs include any adverse event starting on or after the first dose of AMG 820 or pembrolizumab. Relation to study drugs was determined by the investigator. Adverse events (AEs) were graded by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, where Grade 1 = mild AE, Grade 2 = moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening AE, and Grade 5 = death due to AE. Errors in the case report form design resulted in investigators misunderstanding the CTCAE definition for severity grade 5. Therefore data are not reported for severity grade 5. Readers are referred to the 'Fatal TEAE' line in the table below for counts of participants who died during the TEAE timeframe.
Time Frame: Day 1 up to 207 days for Part 1 and Day 1 up to 572 days for Part 2
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 8 | 7 | 41 | 31 | 4 | 19 | 6
Participants
  >=1 TEAE | 8 | 7 | 41 | 31 | 4 | 19 | 6
  Grade >=3 | 7 | 7 | 40 | 30 | 4 | 19 | 6
  Grade >=4 | 2 | 4 | 24 | 26 | 2 | 12 | 4
  Grade >=5 | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning
  Serious AE | 5 | 2 | 31 | 23 | 3 | 11 | 5
  Leading to interruption of AMG 820 | 4 | 3 | 23 | 7 | 1 | 7 | 2
  Leading to discontinuation AMG 820 | 0 | 0 | 6 | 5 | 2 | 1 | 3
  ---- SAE leading to d/c AMG 820 | 0 | 0 | 4 | 4 | 1 | 0 | 2
  ----Non-serious AE leading to d/c AMG 820 | 0 | 0 | 2 | 1 | 1 | 1 | 1
  Leading to discontinuation of PEM | 1 | 0 | 7 | 5 | 2 | 1 | 3
  ---- SAE leading to d/c PEM | 0 | 0 | 4 | 4 | 1 | 0 | 2
  ----Non-serious AE leading to d/c PEM | 1 | 0 | 3 | 1 | 1 | 1 | 1
  Fatal TEAE | 1 | 0 | 4 | 3 | 0 | 3 | 2
  TEAE related to study procedure/activity | 0 | 1 | 11 | 5 | 0 | 3 | 1

3. Primary Outcome: Participants With Treatment -Emergent Adverse Events (TEAEs) Related to AMG 820 Treatment
Description: as for outcome 2
Time Frame: Day 1 up to 207 days for Part 1; Day 1 up to 572 days for Part 2
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 8 | 7 | 41 | 31 | 4 | 19 | 6
Participants
  >=1 TEAE | 5 | 7 | 41 | 25 | 4 | 14 | 6
  Grade >=3 | 3 | 5 | 28 | 11 | 1 | 10 | 6
  Grade >=4 | 1 | 1 | 5 | 5 | 0 | 2 | 2
  Grade >=5 | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning
  Serious AE | 2 | 2 | 12 | 4 | 0 | 3 | 3
  Leading to interruption of AMG 820 | 2 | 3 | 16 | 7 | 0 | 5 | 2
  Leading to discontinuation AMG 820 | 0 | 0 | 3 | 3 | 1 | 0 | 3
  ---- SAE leading to d/c AMG 820 | 0 | 0 | 3 | 2 | 0 | 0 | 2
  ----Non-serious AE leading to d/c AMG 820 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Leading to discontinuation of PEM | 0 | 0 | 4 | 3 | 1 | 0 | 3
  ---- SAE leading to d/c PEM | 0 | 0 | 3 | 2 | 0 | 0 | 2
  ----Non-serious AE leading to d/c PEM | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Fatal TEAE | 0 | 0 | 1 | 0 | 0 | 0 | 1
  TEAE related to study procedure/activity | 0 | 0 | 8 | 2 | 0 | 3 | 1

4. Primary Outcome: Participants With Treatment -Emergent Adverse Events (TEAEs) Related to Pembrolizumab Treatment
Description: as for outcome 2
Time Frame: Day 1 up to 207 days for Part 1 and Day 1 up to 572 days for Part 2
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohort 2: AMG 820 1100 mg + Pem 200 mg | Part 1, Cohort 1: AMG 820 1400 mg + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 8 | 7 | 41 | 31 | 4 | 19 | 6
Participants
  >=1 TEAE | 5 | 7 | 39 | 24 | 4 | 13 | 6
  Grade >=3 | 2 | 5 | 29 | 9 | 1 | 10 | 4
  Grade >=4 | 1 | 1 | 5 | 4 | 0 | 2 | 2
  Grade >=5 | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning | NA — investigator misunderstanding of meaning
  Serious AE | 2 | 2 | 16 | 5 | 0 | 3 | 4
  Leading to interruption of PEM | 1 | 3 | 15 | 6 | 0 | 5 | 2
  Leading to discontinuation AMG 820 | 0 | 0 | 4 | 2 | 1 | 1 | 3
  ---- SAE leading to d/c AMG 820 | 0 | 0 | 3 | 1 | 0 | 0 | 2
  ----Non-serious AE leading to d/c AMG 820 | 0 | 0 | 1 | 1 | 1 | 1 | 1
  Leading to discontinuation of PEM | 0 | 0 | 5 | 2 | 1 | 1 | 3
  ---- SAE leading to d/c PEM | 0 | 0 | 3 | 1 | 0 | 0 | 2
  ----Non-serious AE leading to d/c PEM | 0 | 0 | 2 | 1 | 1 | 1 | 1
  Fatal TEAE | 0 | 0 | 1 | 0 | 0 | 0 | 1
  TEAE related to study procedure/activity | 0 | 0 | 9 | 3 | 0 | 2 | 1

5. Primary Outcome: Objective Response Rate (ORR) Per Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: ORR was defined as the percentage of participants with a best overall response of complete response or partial response assessed by the investigator using immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Response was based on the size of tumors assessed by computed tomography (CT) or magnetic resonance imaging (MRI). During treatment radiographic imaging was performed at Week 10 and repeated at least every 10 weeks until disease progression.
  Complete response (iCR): Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response (iPR): Decrease in tumor burden ≥ 30% relative to baseline. Confirmation by a consecutive assessment at least 4 weeks after first documentation required.
Time Frame: Baseline: Day -28; Treatment: up to Month 13.7
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: AMG 820 + Pem: Part 1 Cohorts 1 + 2 combined. Participants with advanced solid tumors were treated with 1400 mg or 1100 mg AMG 820 plus 200 mg pembrolizumab (Pem) every three weeks (Q3W) to determine safety. Participants could be treated up to 24 months if treatment was tolerable and clinical benefit was observed.
Arm/Group | Part 1: AMG 820 + Pem | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 15 | 41 | 31 | 4 | 19 | 6
percentage of participants | 0.0 [0.00 to 0.00] | 4.9 [0.60 to 16.53] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 5.3 [0.13 to 26.03] | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Time to Response (TTR) Per Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST) For Participants Who Responded
Description: Time to response was defined as the time from first dose of AMG 820 until first documented complete or partial response per irRECIST divided by 365.25 days/12.
Time Frame: Day 1 up to Month 16 (max time to censoring)
Population: Safety Analysis Set
Measure: Mean (Full Range); unit: month
Arm/Group | Part 1: AMG 820 + Pem | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 0 | 2 | 0 | 0 | 1 | 0
month |  | 2.1587 [2.004 to 2.168] |  |  | 2.0698 [NA to NA] — with a single participant contributing data, the full range values equal the observed value. |

7. Secondary Outcome: Time to Progression (TTP) for Participants Who Had Progressive Disease
Description: Time to progression was defined as the time from first dose of AMG 820 until first documented progressive disease per irRECIST divided by 365.25 days/12.
Time Frame: Day 1 up to 14.4 months (max time to censoring)
Population: Safety Analysis Set
Measure: Mean (Full Range); unit: month
Arm/Group | Part 1: AMG 820 + Pem | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 10 | 29 | 13 | 3 | 8 | 4
month | 2.1865 [0.460 to 5.552] | 3.0691 [0.559 to 8.411] | 2.3878 [0.296 to 4.698] | 4.6762 [2.070 to 6.604] | 6.0863 [1.150 to 11.992] | 7.7864 [1.938 to 13.667]

8. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS) at Month 6 and Month 12
Description: Overall survival time was calculated as the number of days from the first administration of AMG 820 to date of death or censoring divided by (365.25/12). Data are reported as the percentage of participants who were alive at Month 6 and Month 12.
Time Frame: Day 1 up to Month 6 or Month 12
Population: Safety Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: AMG 820 + Pem 200 mg: Part 1 Cohorts 1 + 2 combined. Participants with advanced solid tumors were treated with 1400 mg or 1100 mg AMG 820 plus 200 mg pembrolizumab (Pem) every three weeks (Q3W) to determine safety. Participants could be treated up to 24 months if treatment was tolerable and clinical benefit was observed.
Arm/Group | Part 1: AMG 820 + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 15 | 41 | 31 | 4 | 19 | 6
percentage of participants
  Month 6 | 59.077 [32.25 to 78.28] | 53.915 [40.00 to 63.93] | 16.705 [7.40 to 29.24] | 75.000 [22.34 to 94.63] | 52.105 [31.91 to 68.93] | 41.667 [9.26 to 72.47]
  Month 12 | 47.262 [21.19 to 69.63] | 38.963 [25.77 to 51.94] | 8.353 [2.22 to 19.81] | 25.00 [2.08 to 60.89] | 34.737 [17.37 to 52.79] | 41.667 [9.26 to 72.47]

9. Secondary Outcome: Kaplan-Meier Estimates for Progression-Free Survival (PFS) as Per irRECIST at Month 6 and Month 12
Description: Progression-free survival time was calculated as the number of days from the first administration of AMG 820 to date of progressive disease or death or censoring divided by (365.25/12). Data are reported as the percentage of participants who were alive and progression-free at Month 6 and Month 12.
Time Frame: Day 1 up to Month 6 or Month 12
Population: Safety Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: AMG 820 + Pem 200 mg | Part 2, Group 1: CRC MMR-proficient | Part 2, Group 2: Pancreatic Cancer | Part 2, Group 3: NSCLC PD-L1 Low, Naïve | Part 2, Group 4a: Refractory / Relapsing NSCLC PD-L1 Low | Part 2, Group 4b: Refractory/Relapsing NSCLC PD-L1 High
Number analyzed (Participants) | 15 | 41 | 31 | 4 | 19 | 6
percentage of participants
  Month 6 | 10.476 [1.23 to 31.40] | 13.490 [5.99 to 24.04] | 0.000 [0.00 to 0.00] | 25.000 [2.08 to 60.89] | 26.471 [10.67 to 45.41] | 33.333 [7.37 to 62.95]
  Month 12 | 0.000 [0.00 to 0.00] | 5.396 [1.36 to 13.77] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 6.618 [0.77 to 21.97] | 33.333 [7.37 to 62.95]

10. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Time of Maximum Observed Concentration (Tmax) During Treatment Cycles 1 + 2
Time Frame: Cycle 1, Study Day 1: pre-infusion, at end of infusion, hours 1, 6 and 24 post infusion, Days 5, 8 and 15. Cycle 2, Study Day 22: pre-infusion, at end of infusion, hours 1, 6, 24 post infusion, Days 26, 29 and 36
Population: Pharmacovigilence Analysis Set contains all participants who received at least 1 dose of AMG 820 and have at least one PK sample collected.
Measure: Median (Full Range); unit: hour
Groups:
- AMG 820 1100 mg: Includes participants from all treatment arms that were administered AMG 820 1100 mg.
- AMG 820 1400 mg: Includes participants from all treatment arms who were administered AMG 820 1400 mg
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
hour
  Cycle 1 | 2.0 [1.0 to 170] | 2.0 [1.0 to 7.0]
  Cycle 2: number analyzed (Participants) | 71 | 10
  Cycle 2 | 3.00 [1.00 to 25.0] | 2.00 [1.00 to 25.0]

11. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Maximum Observed Drug Concentration (Cmax) During Treatment Cycles 1 + 2
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
ug/mL
  Cycle 1 | 331 (27) | 485 (23)
  Cycle 2: number analyzed (Participants) | 71 | 10
  Cycle 2 | 363 (32) | 536 (21)

12. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Area Under the Curve Last (AUClast) During Treatment Cycles 1 + 2
Description: AUClast is the area under the serum concentration-time curve from time zero to time of last quantifiable concentration.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
hr*ug/mL
  Cycle 1 | 55100 (37) | 80400 (33)
  Cycle 2: number analyzed (Participants) | 71 | 10
  Cycle 2 | 55200 (38) | 73500 (45)

13. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Area Under the Curve Over the Dose Interval (AUCtau) During Treatment Cycles 1 + 2
Description: AUCtau is the area under the serum concentration-time curve over the dose interval tau, with tau equal to 21 days.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
hr*ug/mL
  Cycle 1 | 59300 (33) | 90000 (29)
  Cycle 2: number analyzed (Participants) | 68 | 9
  Cycle 2 | 75400 (35) | 114000 (31)

14. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Minimum Observed Drug Concentration (Cmin) During Treatment Cycles 1 + 2
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
ug/mL
  Cycle 1: number analyzed (Participants) | 70 | 10
  Cycle 1 | 49.9 (51) | 90.9 (35)
  Cycle 2: number analyzed (Participants) | 48 | 3
  Cycle 2 | 78.7 (66) | 199 (34)

15. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Terminal Elimination Half-life (t1/2z) During Treatment Cycles 1 + 2
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
hour
  Cycle 1: number analyzed (Participants) | 46 | 7
  Cycle 1 | 217 (26) | 214 (24)
  Cycle 2: number analyzed (Participants) | 7 | 0
  Cycle 2 | 170 (16) |

16. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Volume of Distribution (Vz) During Treatment Cycles 1 + 2
Description: Volume of distribution observed at terminal phase after intravenous dosing.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
liter
  Cycle 1: number analyzed (Participants) | 46 | 7
  Cycle 1 | 5200 (35) | 4110 (25)
  Cycle 2: number analyzed (Participants) | 7 | 0
  Cycle 2 | 4560 (21) |

17. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Drug Clearance (CL) During Treatment Cycles 1 + 2
Description: Drug clearance observed after intravenous dosing.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
liter/hour
  Cycle 1: number analyzed (Participants) | 46 | 7
  Cycle 1 | 16.6 (37) | 13.3 (33)
  Cycle 2: number analyzed (Participants) | 7 | 0
  Cycle 2 | 18.6 (30) |

18. Secondary Outcome: AMG 820 Pharmacokinetic Parameter by Dose Group: Accumulation Ratio (AR)
Description: Accumulation ratio is AUCtau following administration in Cycle 2 / AUCtau after administration in Cycle 1
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AMG 820 1100 mg | AMG 820 1400 mg
Number analyzed (Participants) | 97 | 18
ratio | 1.23 (18) | 1.25 (16)

ADVERSE EVENTS:
Time Frame: The TEAE timeframe was Day 1 up to 207 days for Part 1 and Day 1 up to 572 days for Part 2. The median time frame is 122 days.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All adverse events (AEs) and disease related events (DREs) are integrated in above summaries.
Groups:
- AMG 820 1400 MG: Includes participants from all treatment arms that were administered AMG 820 1400 mg.
Arm/Group | AMG 820 1100 MG | AMG 820 1400 MG
All-Cause Mortality (participants affected / at risk) | 12/98 | 1/18
Serious Adverse Events (participants affected / at risk) | 70/98 | 10/18
Other Adverse Events (participants affected / at risk) | 97/98 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 820 1100 MG (N=98) | AMG 820 1400 MG (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 3 | 0
Fatigue (General disorders) | 2 | 2
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 3 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 3 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 0
Urosepsis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 820 1100 MG (N=98) | AMG 820 1400 MG (N=18)
Anaemia (Blood and lymphatic system disorders) | 35 | 4
Bradycardia (Cardiac disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 6 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 38 | 10
Periorbital swelling (Eye disorders) | 2 | 1
Photophobia (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 2
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 20 | 6
Ascites (Gastrointestinal disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 22 | 9
Diarrhoea (Gastrointestinal disorders) | 23 | 5
Dry mouth (Gastrointestinal disorders) | 8 | 3
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 26 | 7
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 12 | 5
Asthenia (General disorders) | 8 | 0
Chills (General disorders) | 11 | 3
Face oedema (General disorders) | 14 | 5
Fatigue (General disorders) | 52 | 10
Hyperthermia malignant (General disorders) | 0 | 1
Oedema (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 10 | 2
Pain (General disorders) | 6 | 0
Pyrexia (General disorders) | 25 | 3
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 8 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 1
Mucosal infection (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 5 | 0
Skin infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 6 | 0
Viral infection (Infections and infestations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 6 | 0
Alanine aminotransferase (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 21 | 4
Amylase increased (Investigations) | 19 | 5
Aspartate aminotransferase abnormal (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 58 | 12
Blood alkaline phosphatase increased (Investigations) | 13 | 5
Blood bilirubin increased (Investigations) | 5 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 5 | 0
Lipase increased (Investigations) | 18 | 5
Liver function test abnormal (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 7 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 6 | 1
White blood cell count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 22 | 9
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 18 | 8
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 4
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 5 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 2
Lethargy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 2
Confusional state (Psychiatric disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 4 | 4
Bladder spasm (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 7 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 4
Rash (Skin and subcutaneous tissue disorders) | 25 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 16 | 4
Hypotension (Vascular disorders) | 5 | 0
Venous thrombosis (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT02713529/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02713529/SAP_001.pdf